CLINICAL TRIAL: NCT03379896
Title: Study on Antigen-presenting Function of Gamma Delta T Cells in Sepsis and Its Molecular Mechanisms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, Yan Kang, Director of Department of Critical Care Medicine, West China Hospital
Other Study IDs: 81701880
Record Dates: First submitted 2017-12-16; First posted 2017-12-20 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Sepsis; Antigen-presenting Function; γδ T Cells
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: Patient diagnosed with sepsis according to the new sepsis definition (infection+SOFA≥2).
  Interventions: Other: Collect peripheral blood sample
- Control: Age-matched healthy control
  Interventions: Other: Collect peripheral blood sample

INTERVENTIONS:
Other: Collect peripheral blood sample — Collect 20 ml heparinized blood from patients and controls strictly abiding by the principle of aseptic manipulation after informed consent.

SUMMARY:
Study on antigen-presenting function of gamma delta T cells in sepsis and its molecular mechanisms

DETAILED DESCRIPTION:
The latest definition of sepsis highlights the role of dysregulated host response to infection in organ dysfunction aggravation. Maintenance of immune homeostasis of septic patients through immunotherapy is the key breakthrough to improve success rate. Antigen-presenting cell (APC) is the bridge that connects the innate and adaptive immunity. Decrease of count and function of APC has been shown to be associated with worsened clinical outcomes in patients with sepsis. Gamma-delta T cells (γδ T cells) are the newly identified population of T lymphocytes. Recent studies have found that γδ T cells possess unique and powerful antigen-presenting function, making them the hot topic in infection and cancer research. Based on the results, the investigator plan to evaluate the antigen-presenting function changes of γδ T cells in septic status by analyzing the antigen-presenting related molecules on γδ T cells, antigen protein uptake ability, and their function on the proliferation and activation of CD8+ T lymphocytes. Furthermore, the investigator will explore the mechanism and signal pathways for the APC function changes of γδ T cells. Findings from this research could help explain the mechanism of sepsis induced immune dysfunction, enrich our understanding of the important role of γδ T cells, and build a good foundation for immunotherapy in sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 year old;
2. a known or suspected infection based on clinical data at the time of admission and sepsis-induced dysfunction of at least one organ.

Exclusion Criteria:

1. autoimmune disease,
2. history of transplantation,
3. acute tuberculosis,
4. chronic hepatitis B or C infection,
5. HIV infection,
6. active malignancy, and
7. long-term use of cortical steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis from department of Critical Care Medicine of West China Hospital are included if they meet the study criteria on ICU admission. Healthy control subjects are adult volunteers from our hospital staff and their family members with no significant acute or chronic illnesses.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-04 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
28-day clinical outcome | 28-day after ICU admission
  death

IPD SHARING:
Plan to Share IPD: Undecided